CLINICAL TRIAL: NCT05362825
Title: Surgery Outcome Treated by Neo-adjuvant Chemotherapy FOLFOXIRI Regimen in Colorectal Cancer With Liver-limited Synchronous Metastases
Brief Title: Surgery Outcome Treated by Neo-adjuvant Combination of Oxaliplatin, Irinotecan, Folinic Acid and Fluorouracil (FOLFOXIRI) Regimen in Synchronous Liver Limited Metastasis Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cho Ray Hospital (Other)
Collaborators: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Vuong Dinh Thy Hao, Doctor, Medical Oncologist, Cho Ray Hospital at Ho Chi Minh City, Cho Ray Hospital
Other Study IDs: Cho Ray hospital
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Liver Metastasis Colon Cancer; Synchronous Neoplasm
Keywords: FOLFOXIRI
MeSH Terms: conditions — Neoplasms, Multiple Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Un-resectable synchronous liver limited metastasis colorectal cancer: Un-resectable synchronous liver limited metastasis colorectal cancer patients undergoing neo-adjuvant chemotherapy FOLFOXIRI regimen, up to 12 cycles.
  Interventions: Drug: Neo-adjuvant Chemotherapy FOLFOXIRI Regimen; Procedure: synchronous resection surgery

INTERVENTIONS:
Drug: Neo-adjuvant Chemotherapy FOLFOXIRI Regimen — Oxaliplatin 85mg/m2 IV; Irrinotecan 165mg/m2 IV; Leucovorin 400mg/m2 IV; 5-Fluorouracil 2400mg/m2 continuous infusion in 46 hours - every 2-week cycle, up to 12 cycles.
Procedure: synchronous resection surgery — Patients undergoing colorectal primary and liver resection in a single operation or staged curative procedure or no surgery
  Other Names: Liver-first surgery; Primary/Bowel-first Surgery; No surgery

SUMMARY:
This single arm study aims to evaluate the rate of conversion therapy in patients with unresectable liver-limited metastatic colorectal cancer (mCRC) using FOLFOXIRI neoadjuvant regimen and to assess the other outcome including the response rate, the survival rate and the safety profile.

DETAILED DESCRIPTION:
Patients with liver-only metastases colorectal cancer could potentially be cured following surgical resection of metastases. Recent evidence suggest that a triplet chemotherapy regimen, FOLFOXIRI has been associated with higher R0 resection.

Eighty-nine eligible patients will be recruited at Cho Ray hospital in Vietnam. Patients will receive neoadjuvant FOLFOXIRI regimen every two weeks for up to 12 cycles and will undergo periodic imaging studies. The resectability of liver metastases will be assessed by a multidisciplinary team comprised of digestive surgeons, hepato-biliary surgeons, radiologists, and oncologists. This study will be helpful to establish a standard chemotherapy regimen for patients with liver-limited metastatic colorectal cancer. Moreover, this study will assess the surgical outcome, the response rate, the survival rate, the safety of triple drug chemotherapy and the association between conversion operable disease and various survival rate and patient's characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 75 years
* Able to give informed consent
* Have a histological adenocarcinoma diagnosis of colorectal cancer
* Resected or operable colorectal primary tumor
* Initially unresectable liver lesion considered by multidisciplinary team (MDT)
* World Health Organisation performance status (ECOG PS) 0, 1
* Adequate complete blood count, liver and renal function

Exclusion Criteria:

* Prior history of other active malignancies
* Unmeasurable lesion according to RECIST criteria v.1.1
* Recurrence of colorectal cancer
* Resection or ablation of liver lesion
* Distant metastases outside the liver
* Patients who have received prior chemotherapy with Oxaliplatin, Irinotecan, Capecitabine, 5-Fluoro-uracil.
* Concomitant uncontrollable medical status ie. symptomatic cardiac disease, infarction within 24 months, uncontrollable cardiac dysrhythmia, active infectious disease
* Pathology of the liver lesion except adenocarcinoma metastasis from colorectal cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise patients with colorectal cancer with un-resectable synchronous liver-limited hepatic metastases
Sampling Method: Non-Probability Sample
Enrollment: 89 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-01-23 (Estimated)

PRIMARY OUTCOMES:
Resectable outcome | 8 weeks
  R0 resection rate of liver metastases; Intra operative accident; Post-operative accident

SECONDARY OUTCOMES:
Progression free survival | 5 years
Overall survival | 5 years
The incidence of chemotherapy related adverse events | 2 weeks
  Incidence of the adverse events in any grade; the serious adverse events

OTHER OUTCOMES:
Correlation between R0 procedure and patient's characteristics. | 8 weeks
  age, sex, ECOG PS, colon site, Carcinoembryonic antigen (CEA) level, RAS/ BRAF gene mutation, chemotherapy cycle numbers, Early tumor shrinkage; Depth of response; Surgery procedure; Liver lesion's number; Liver lesion's site, Liver lesion's dimension
Correlation between R0 procedure and survival time | 5 years
  Progression free survival (PFS) time, Overall survival (OS) time

CONTACTS AND LOCATIONS:
Locations (1):
- Cho Ray hospital- 201 B Nguyen Chi Thanh, District 5, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Siriwardena AK, Mason JM, Mullamitha S, Hancock HC, Jegatheeswaran S. Management of colorectal cancer presenting with synchronous liver metastases. Nat Rev Clin Oncol. 2014 Aug;11(8):446-59. doi: 10.1038/nrclinonc.2014.90. Epub 2014 Jun 3. PMID 24889770
- [Result] Masi G, Allegrini G, Cupini S, Marcucci L, Cerri E, Brunetti I, Fontana E, Ricci S, Andreuccetti M, Falcone A. First-line treatment of metastatic colorectal cancer with irinotecan, oxaliplatin and 5-fluorouracil/leucovorin (FOLFOXIRI): results of a phase II study with a simplified biweekly schedule. Ann Oncol. 2004 Dec;15(12):1766-72. doi: 10.1093/annonc/mdh470. PMID 15550581
- [Result] Souglakos J, Androulakis N, Syrigos K, Polyzos A, Ziras N, Athanasiadis A, Kakolyris S, Tsousis S, Kouroussis Ch, Vamvakas L, Kalykaki A, Samonis G, Mavroudis D, Georgoulias V. FOLFOXIRI (folinic acid, 5-fluorouracil, oxaliplatin and irinotecan) vs FOLFIRI (folinic acid, 5-fluorouracil and irinotecan) as first-line treatment in metastatic colorectal cancer (MCC): a multicentre randomised phase III trial from the Hellenic Oncology Research Group (HORG). Br J Cancer. 2006 Mar 27;94(6):798-805. doi: 10.1038/sj.bjc.6603011. PMID 16508637
- [Result] Marques RP, Duarte GS, Sterrantino C, Pais HL, Quintela A, Martins AP, Costa J. Triplet (FOLFOXIRI) versus doublet (FOLFOX or FOLFIRI) backbone chemotherapy as first-line treatment of metastatic colorectal cancer: A systematic review and meta-analysis. Crit Rev Oncol Hematol. 2017 Oct;118:54-62. doi: 10.1016/j.critrevonc.2017.08.006. Epub 2017 Aug 25. PMID 28917269
- [Derived] Hao VDT, Tri PM, My DT, Anh LT, Trung LV, Bac NH, Vuong NL. FOLFOXIRI for First-Line Treatment of Unresectable Colorectal Cancer with Liver Metastases in a Resource-Limited Setting. J Gastrointest Cancer. 2024 Oct 31;56(1):12. doi: 10.1007/s12029-024-01133-4. PMID 39480530